CLINICAL TRIAL: NCT06324617
Title: Treatment of Failed Carpal Tunnel Syndrome by Dorsal Ulnar Artery Perforator Adipofascial Flap
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Shehata Gaber, specialist of Orthopaedics Orthopaedic and Traumatology department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-Med-24-02-06MS
Record Dates: First submitted 2024-03-10; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Failed Carpal Tunnel Syndrome Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Treatment of failed carpal tunnel syndrome by dorsal ulnar artery perforator adipofascial flap — Treatment of failed carpal tunnel syndrome by dorsal ulnar artery perforator adipofascial flap The previous incision is reopened and extended, Neurolysis begins proximally preserving the palmar cutaneous branch. The subcutaneous tissue is exposed, leaving part of the superficial venous plexus with the adipofascial flap. Flap elevation is begun by incising the subcutaneous tissue through the deep fascia along the radial border of FCU and ECU .
  When the flap reaches a suitable length (10-12 cm from the wrist), it is cut proximally and along the ulnar side. The flap is dissected proximally to distally in continuity with the underlying fascia . When the dissected flap is (2-5) cm proximal to the wrist. Ulnar retraction of the flexor carpi ulnaris permits identification of the perforator. the pivot point of the flap is localized (2-5) cm proximal to the pisiform.
  The adipofascial flap is turned 180 degrees and anchored with a few absorbable stitches around the median nerve.

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common compressive neuropathy in the general population. Surgical treatment by open or endoscopic carpal tunnel release (CTR) is the first choice of treatment and has clinical success rates of 75% to 90%.The rate of recurrence after primary median nerve release is 3-19% [1,2]. Between 0.3% and 12% of cases require surgical revision [2,3]. The risk factors for surgical revision for secondary release are male gender, staged or simultaneous bilateral carpal tunnel release, endoscopic release, smoking and rheumatoid arthritis.

Treatment failures after primary CTR are classified as persistent CTS, recurrent CTS, or new symptoms. Recurrent symptoms are uncommon and are defined by a symptom-free interval after surgery. Persistent symptoms are relatively common, particularly in elderly patients and in patients with concurrent nerve compression or medical conditions that affect nerve function, such as diabetes. Persistent or recurrent CTS principally results from incomplete release of the transverse carpal ligament but may be accompanied by perineural scarring, leading to compression or tethering of the median nerve.

New symptoms may be caused by iatrogenic nerve injury. Surgical treatment of recurrent or persistent CTS after primary CTR usually involves open revision CTR, extended proximally into unscarred tissue, and has also included internal or external neurolysis. Unsatisfactory results following revision CTR are common.

A second compression site, or double-crush syndrome, may clinically present as RCTS or PCTS . Thorough preoperative clinical examination may uncover signs of a second compression site, which can then be confirmed on electroneuromyography (ENMG) of the entire arm.

To improve outcomes of revision CTR, recent studies have emphasized the importance of median nerve coverage by well-vascularized soft tissue to enhance nerve healing, to prevent tethering in surrounding scar tissue, and to optimize nerve gliding in the carpal tunnel. Several local flaps (hypothenar fat pad flap, tenosynovial flap), regional flaps (posterior interosseous artery flap, reverse radial artery fascial flap, flexor digitorum superficialis flap), and free flap techniques have been described, but consensus for specific flap has not been reached. Following potential iatrogenic median nerve injury and reexploration for a painful neuroma incontinuity, flap coverage may also be beneficial.

In 1988, Becker and Gilbert introduced a Fasciocutaneous pedicled flap based on a consistent dorsal perforator of the ulnar artery (absent in 1 % of population) named the dorsal ulnar artery (DUA) flap or simply the Becker flap. The authors described open revision CTR with nerve coverage by a DUA flap in 3 patients with recurrent CTS and reported good results as well as a quick and easy-to-perform dissection with low donor site morbidity and preservation of the radial andulnar artery. Since this introduction, additional studies describing fasciocutaneous DUA flaps have mostly focused on its use for reconstruction of hand or wrist wounds. Despite the original described benefits, additional studies of DUA flaps for the treatment of recurrent or persistent CTS have remained limited.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Positive tinel sign
* Operative interval more than 3 months & less than 2 years

Exclusion Criteria:

* Cervical disc
* Associated general disease (Rheumatoid arthritis, DM ,psychological problems & peripheral neuropathy)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain visual analogue scale (VAS) | 1 year
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end .meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels.Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain".the position of the respondent's cross is generally assigned a score between 0 and 100. If documented in paper form, the scores can then be simply transferred to a 100-value scale using a millimeter tape measure

SECONDARY OUTCOMES:
Two point discrimination test | 1 year
  one of the most commonly used neurosensory tests to assess mechanoperception in the clinical settings. While there have been numerous studies of functional sensibility of the hand using TPD test.
Tinel sign | 1 year
  a tingling or "pins and needles" feeling you get when your healthcare provider taps your skin over a nerve. Tinel's sign may be an indicator that you have nerve compression or damage where they're tapping

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bollmann G, Bouvet C, Beaulieu JY. Recurrent carpal tunnel syndrome: Outcomes after neurolysis and synovial flap. Hand Surg Rehabil. 2023 Jun;42(3):236-242. doi: 10.1016/j.hansur.2023.04.004. Epub 2023 Apr 25. PMID 37105520
- [Background] Neuhaus V, Christoforou D, Cheriyan T, Mudgal CS. Evaluation and treatment of failed carpal tunnel release. Orthop Clin North Am. 2012 Oct;43(4):439-47. doi: 10.1016/j.ocl.2012.07.013. Epub 2012 Aug 30. PMID 23026459
- [Background] Lauder A, Mithani S, Leversedge FJ. Management of Recalcitrant Carpal Tunnel Syndrome. J Am Acad Orthop Surg. 2019 Aug 1;27(15):551-562. doi: 10.5435/JAAOS-D-18-00004. PMID 30973521
- [Background] Botte MJ, von Schroeder HP, Abrams RA, Gellman H. Recurrent carpal tunnel syndrome. Hand Clin. 1996 Nov;12(4):731-43. PMID 8953292